CLINICAL TRIAL: NCT05197881
Title: Daily Adaptive External Beam Radiation Therapy in the Treatment of Carcinoma of the Cervix: A Prospective Trial of an Individualized Approach for Intestinal Toxicity Reduction (ARTIA-Cervix)
Brief Title: Daily Adaptive Radiation Therapy an Individualized Approach for Carcinoma of the Cervix
Acronym: ARTIA-Cervix
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-04
Record Dates: First submitted 2021-11-30; First posted 2022-01-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer by FIGO Stage 2018

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Daily Adaptive External Beam Radiation Therapy (Experimental): Daily adaptive radiation therapy delivered with Varian Ethos treatment system.
  Interventions: Device: Varian Ethos Adaptive Radiation Therapy

INTERVENTIONS:
Device: Varian Ethos Adaptive Radiation Therapy — Daily adaptive external beam radiation therapy delivered on Varian Ethos treatment system.

SUMMARY:
This is a single-arm, prospective, multi-center clinical trial designed to demonstrate that adaptive radiotherapy for locally advanced cervical cancer will translate into a decreased rate of acute gastrointestinal toxicity compared with the historically reported rate for non-adaptive intensity modulated radiation therapy (IMRT). The timepoint for this assessment will be at week 5 of external beam radiotherapy (EBRT) and will use the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed, newly diagnosed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma): FIGO 2018 clinical stages IB2-IVA, without involved paraaortic lymph nodes.
2. For patients with involved pelvic lymph nodes, the upper border of the CTV nodal volume may not extend above the confluence of the common iliac arteries with the aorta (i.e., aortic bifurcation).
3. Patients must NOT have had a hysterectomy.
4. Pelvic nodal status is to be confirmed by one or more of the following studies/procedures: PET/CT scan, CT scan, MR Scan, fine needle biopsy, extra peritoneal biopsy or laparoscopic biopsy, per institutional standard of care.
5. Patients must be planning to undergo concurrent pelvic radiation and chemotherapy.
6. ECOG performance status ≤ 2 (Karnofsky ≥60%).
7. Patient must be willing and able to complete the PRO-CTCAE, EQ-5D, EPIC and EORTC questionnaires as described in the study protocol.
8. Patient must have normal organ and marrow function as defined below:

   * leukocytes ≥ 2,500/mcL
   * absolute neutrophil count ≥ 1,500/mcL
   * platelets ≥ 100,000/mcL
   * hemoglobin ≥ 8 g/dL (can be transfused with red blood cells pre-study)
   * total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
   * AST(SGOT)/ALT(SGPT) ≤ 3 × ULN
   * alkaline phosphatase ≤ 2.5 × ULN
   * creatinine < 1.5 mg/dL to receive weekly cisplatin*

     * Patients whose serum creatinine is between 1.5 and 1.9 mg/dL are eligible for cisplatin if there is no hydronephrosis and the estimated creatinine clearance (CCr) is >30 ml/min. For the purpose of estimating the CCr, the formula of Cockcroft and Gault for females should be used:CCr=(0.85 ×(140-age)×IBW)/((Scr×72)) where age is the patient's age in years (from 20 to 80 years), Scr is the serum creatinine in mg/dL, and IBW is the ideal body weight in kg (according to the calculation IBW = 45.5 kg + 2.3 kg for each inch over 5 feet).
9. Age ≥ 18 years (or meets local age of consent).
10. Study participant is already intending to be prescribed a standard of care cisplatin treatment regimen.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior radiation therapy to the pelvis or abdominal cavity, para-aortic lymph glands (PALN) radiation, or previous therapy of any kind for this malignancy.
2. Patients with PALN nodal metastasis.
3. Patients who have undergone staging pelvic and/or paraaortic lymphadenectomy.
4. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
5. Prior systemic anticancer therapy due to a diagnosis of cancer (e.g., chemotherapy, targeted therapy, immunotherapy) within 3 years prior to entering the study.
6. Patients diagnosed on imaging or biopsy with a synchronous primary malignancy (with the exception of DCIS of the breast, or early stage basal cell carcinoma of the skin).
7. Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease.
8. Patients with a history of other symptomatic autoimmune disease: rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's Granulomatosis); CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis, multiple sclerosis.).
9. Patients with active tuberculosis (TB).
10. Patients who are pregnant.
11. Patients who are actively breastfeeding (or who do not agree to discontinue breastfeeding before the initiation of protocol therapy).
12. Patients who are of child-bearing potential who do not agree to use birth control (for a minimum of 14 months after the last dose of cisplatin) in accordance with institution's standard of care.
13. Patients with a prior known history or current diagnosis of a vesicovaginal, enterovaginal, or colovaginal fistula.
14. Patients who undergo a pelvic or para-aortic lymph node dissection prior to planned chemoradiation therapy.
15. Patients with known active infection of HIV.
16. Patients with hip prosthetics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Acute Patient Reported Outcome (PRO) GI Toxicity | End of external beam treatment delivery (week 5)
  GI toxicity as reported by the patient using the gastrointestinal section of the NCI-PRO questionnaire

SECONDARY OUTCOMES:
Key powered secondary endpoint: Fecal Urgency | End of external beam treatment delivery (week 5)
  Acute reported fecal urgency (as measured by the inability to defer defecation by 15 minutes)
Acute PRO Bowel Toxicity | End of external beam treatment delivery (week 5)
  Bowel toxicity as reported with EPIC bowel questionnaire
Acute PRO Urinary Toxicity | End of external beam treatment delivery (week 5)
  Urinary toxicity as reported with EPIC urinary questionnaire
Patient Reported Quality by EQ-5D-5L | 24 months post treatment
  Quality of life as document with EQ-5D-5L patient reported questionnaire
Patient Reported Quality by EORTC | 24 months post treatment
  Quality of life as document with EORTC patient reported questionnaire
Disease-free Survival | Enrollment through 2 year follow up
  Disease-free survival at 2 years
Normal Tissue Complication Probability Model | Enrollment through 2 year follow up
  Develop a normal tissue complication probability (NTCP) model of acute GI toxicity based on true integrated daily dose to the bowel
Workflow Feasibility | End of external beam treatment delivery
  Record percentage of fractions delivered with adaptive radiation therapy vs traditional IGRT
CTCAE Toxicities | Enrollment through 2 year follow up
  Physician reported CTCAE toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mayadev, MD, Principal Investigator — University of California, San Diego; Xenia Ray, PhD, Principal Investigator — University of California, San Diego
Locations (5):
- United States (5):
  - University of Alabama Birmingham, Burmingham, Alabama
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No